CLINICAL TRIAL: NCT06178107
Title: UOC DI GASTROENTEROLOGIA AOU S.GIOVANNI DI DIO E RUGGI D'ARAGONA (Italy) & University of Roehampton (UK)
Brief Title: Efficacy of Cholesterol-lowering L. Plantarum on Cardiometabolic Health Biomarkers in Coeliac Disease Patients
Acronym: ProCoChoL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Study PI, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LSC 23/ 395
Record Dates: First submitted 2023-11-17; First posted 2023-12-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Celiac Disease
Keywords: PROBIOTICS, HIGH CHOLESTEROLEMIA
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: This is a double blinded, randomised of parallel design pilot study will include 50 adults aged 18-65 with coeliac disease (CD). After an initial screening, potential subjects will be assessed for inclusion in the run-in trial.
  Those subjects who meet the inclusion criteria will be then invited to the intervention study for a total duration of 9 weeks, followed by 3 weeks follow up.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus plantarum (LPLDL®) equivalent to 4 x10^9 CFU (0.1 g) with the addition of filling carrier (0.12 g; 30% w/v maltodextrin and 5% w/v sucrose) as a capsular format (vegetable) to be consumed once a day, after lunch with 250mL of water.
  Interventions: Dietary Supplement: LP-LDL Probiotic
- placebo (Placebo Comparator): Maltodextrin (an oligosaccharide without prebiotic effect) (0.12 g; 30% w/v maltodextrin and 5% w/v sucrose) as a capsular format (vegetable) to be consumed once a day, after lunch with 250mL of water.
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: LP-LDL Probiotic — LP-LDL a dietary food supplement probiotic
  Other Names: Placebo Comparator
  Arms: Probiotic
Dietary Supplement: Placebo Comparator — Placebo comparator Maltodextrin
  Arms: placebo

SUMMARY:
Recent studies have also shown that 30% of the world's population carries the susceptibility genes for coeliac disease and that only 2-5% of these individuals are really affected, however, studies suggest the existence of other factors capable of contributing to the onset of the disease, such as intestinal dysbiosis. We have also seen how each of us has a specific microbiota, defined as an individual human enterotype, which depends on our background and can be modified by the diet. Recently, much interest has been directed to a strain of lactobacilli, called Lactobacillus plantarum (LP-LDL®) capable of reducing cholesterol and preventing the reabsorption of bile salts in the liver. The efficacy of this bacterial strain has been confirmed in 3 different human studies demonstrating the efficacy of LP-LDL® in patients with high baseline cholesterol (TC> 6mmol / L). This is a food supplement that has been commercially available in multiple formulations in Europe for over 3 years. LP-LDP is a probiotic strain, safe to use, selected for its high bile salt hydrolase in vitro, and in vivo cholesterol reduction activity. The intake of 2 Å~ 109 CFU encapsulated LP-LDL twice daily, significantly reduced LDL-C (13.9%), total cholesterol (TC) (37.6%), TG (53.9%), and significantly increased HDL-C (14.7%; in subjects >60 years of age; 6-12 weeks) in normal to mildly hypercholesterolaemic subjects. In a recent double-blind placebo-controlled human study published by the Journal of Functional Foods (2022) and carried out by the University of Roehampton (UK), LPLDL showcased statistically significant reductions in multiple cardiovascular risk biomarkers, including total cholesterol, LDL cholesterol, non-HDL cholesterol and apoB. No adverse effects were noted throughout the study.

We are here proposing a pilot human intervention study to evaluate the effectiveness of the LP-LDL® probiotic in reducing cardiovascular risk factors inclusive of cholesterol in the blood in people with coeliac disease.

DETAILED DESCRIPTION:
A total of 50 coeliac subjects (+/- 6 additional volunteers) will be recruited to achieve statistical significance with changes on a logarithmic scale of 1.2 for cholesterol based on other interventional studies using focused probiotics on the reduction of the lipid picture. Based on these calculations, 10 coeliac subjects are required for each study group. The Mann-Whitney U test will be used to compare variables that are not normally distributed. GraphPad Prism Version 9.0 (GraphPad Software, Inc., San Diego, CA, USA) will be used for statistical analysis. All patients with coeliac disease will be recruited at Roehampton until the set target by the Protocol (at least 25 patients will be enrolled). This is to ensure we have an acceptable number of patients that can be monitored, net of subjects lost to follow up (drop-out). A random generator (GraphPad QuickCalcs, San Diego, CA, USA) will be used in order to assign a specific number to each patient and ensure double-blind randomization of the 50 patients in two study groups. Patients will be stratified by gender and randomly assigned to one of the two treatment groups using a 2: 1 ratio due to the higher prevalence of female sex in coeliac patients.

ELIGIBILITY:
Inclusion criteria

* Adults aged between 18 and 65 years, with CD Diagnosis
* Fasting blood glucose level not above 5.6-6.9mmol/L
* High baseline cholesterol (TC> 6mmol / L).
* HbA1c below 5.7%
* With cholesterol
* For intervention purposes, eligible participants are also required to have a mobile phone and be able to read and speak English.

Exclusion criteria

* People with comorbid conditions that may limit participation in the study, such as a history of an acute cardiovascular event, uncontrolled hypertension, cancer or major psychiatric or cognitive problems
* People who are already participating in a weight loss programme
* People receiving drug treatment for lipid metabolisms (e.g., statins
* People with a history of long-term use of medicines known to influence glucose metabolism (e.g., corticosteroids)
* People with elevated liver enzymes (alanine aminotransferase ≥300 IU/L, aspartate aminotransferase ≥300 IU/L)
* People who take antibiotics or bacterial agents (Probiotics) within 1 month
* Pregnant women, women ready for pregnancy, and nursing mothers

All capsules (probiotic and placebo) have the same taste and appearance and have been mixed, encapsulated and packaged to ensure product consistency throughout the study. All capsules will be distributed free of charge to participants in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in blood cholesterol levels | Change from baseline to 6 and 9 weeks of the intervention
  To test, in humans, whether LPLDL® intervention lowers total cholesterol compared to the baseline levels
Change in BMI (body mass index) Scores | Change from baseline to 6 and 9 weeks of the intervention
  To test wheter LPLDL® intervention affect body mass indes in kg/m^2

SECONDARY OUTCOMES:
Change in the gut microbiota diversity | Change from baseline to 6 and 9 weeks of the intervention
  To determine the effect of LPLDL® on the faecal microbiota composition and microbial composition express as ratio compared to the baseline levels
Change in dietary habits | Change from baseline to 6 and 9 weeks of the intervention
  To conduct an assessment of dietary intake in the study population using a validated four-day food diary compared to the baseline levels
Change in VitD levels | Change from baseline to 6 and 9 weeks of the intervention
  To determine the effect of LPLDL® in VITD profile express in mmol/L compared to the baseline
Change in ApoB concentration | Change from baseline to 6 and 9 weeks of the intervention
  To determine the effect of LPLDL® in ApoB levels express in mmol/L in comparison to baseline levels

CONTACTS AND LOCATIONS:
Overall Officials: Adele Costabile, Prof, Study Director — Roehampton University
Locations (2):
- Uoc Di Gastroenterologia Aou S. Giovanni Di Dio E Ruggi D'Aragona, Salerno, Italy
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No